CLINICAL TRIAL: NCT05920577
Title: Effects of the Combined Use of Exergaming and Resistance Training in Improving the Frailty of Nursing Home Residents: A Pilot Randomised Controlled Trial
Brief Title: Effects of Exergames and Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Liu Tai Wa, Associate Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Frailty_2023
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Frailty; Sacropenia; Cognition; Mood; Mobility
Keywords: Nursing home residents; Frailty; Sacropenia
MeSH Terms: conditions — Frailty | interventions — Exergaming; Resistance Training

STUDY DESIGN:
Intervention Model Description: This pilot randomised controlled trial will conduct in a nursing home starting from Aug 2023 in Hong Kong
Who Masked: Outcomes Assessor
Masking Description: After the baseline assessment, all eligible participants will be allocated randomly in a 1:1 ratio to either (1) experimental group which received exergaming and resistance training over a period of 12 weeks, or (2) control group which received resistance training over a period of 12 weeks. The research assistant, who is responsible for allocation, is independent from the data collection and anslysis, and the intervention. The participants will be reminded not to disclose information related to group allocation to the assessors to prevent possible bias during measurement. All assessments will be performed by an assessor who is blinded to the group allocation and not involved in the delivery of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exergames and resistance training group (Experimental): Participants will receive exergaming and resistance training programme over a period of 12 weeks
  Interventions: Other: exergames and resistance training
- Resistance training group (Active Comparator): Participants will receive resistance training programme over a period of 12 weeks
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: exergames and resistance training — In each session, the participants will receive 40 minutes of combined use of exergaming and resistance training. The participants will practice the exergames using the gaming system Nintendo Switch (Nintendo Co., Ltd, Kyoto, Japan). The gaming software "Nintendo Switch Sports" will be adopted in which arrays of exergames are available to strengthen both the upper and lower extremity muscle and improve the balance ability of participants. The exergaming programme will consist of both upper (badminton game and tennis game) and lower (soccer game) extremity games. For week 1 and 2, the participants will first practice 1-minute warm up exercise (stretching exercises) and then the 3 exergames. For week 3 to 12, the participants will receive the same warm up exercise and exergames as if week 1 and 2 but there will be an addition of light cuff weight for resistance training.
  Arms: Exergames and resistance training group
Other: Resistance training — The resistance training programme consists of 2 parts, the upper limb and lower limb resistance exercises. For the upper limb resistance exercises, the participants will first practice 5-minute warm up of upper limb using ergometer and then undergo 2 resistance exercises, including handgrip and elbow flexion. For the lower limb exercise, the participants will also first practice 5-minute warm up of lower limb using ergometer and then undergo 3 resistance exercises, including squatting, single-leg standing and knee extension.
  Arms: Resistance training group

SUMMARY:
Frailty is a common geriatric condition with significantly increased vulnerability to stress and susceptibility of negative health-related outcomes. Sacropenia and impaired cognitive function are two major contributors to frailty. This study aims to evaluate the effects of the combined use of exergaming and resistance training in improving the frailty of nursing home residents.

DETAILED DESCRIPTION:
Frailty is a common geriatric condition with significantly increased vulnerability to stress and susceptibility of negative health-related outcomes. The prevalence rates of frailty varies across countries, and the pooled estimates of prevalence rates of 52.3% and 40.2% of frailty and prefrailty were reported among nursing home residents respectively. Previous studies also revealed that frailty is predictive for various adverse health outcomes.

Sacropenia is a major etiologic risk factor to frailty. It refers to an age-related generalised muscle disorder featuring with loss of muscle mass and function5. Talar et al systematically reviewed and meta-analysed 25 randomised controlled trials (RCTs) using resistance training among 2,267 older people (age >65 years) with pre-sarcopenia, sarcopenia, pre-frailty or frailty. It was revealed that, compared to control, resistance training with at least 8 weeks intervention period had small to large effects in improving handgrip strength, lower-limb strength, agility, gait speed, postural stability, functional performance, fat mass and muscle [Effect size (ES) = 0.29 - 0.93, p <0.001 to = 0.007].

Cognitive impairment is another major risk factor for declined frailty status among prefrail older people. Non-frail older people are known to have better performance on cognitive status, including processing speed, executive function, attention and working memory, immediate memory and delayed memory (g = 0.320 to 0.64), than frail older people. Ample research evidence suggested that cognition predicts the incidence of frailty.

Exergaming is a fast growing research trend in gerontechnology and several commercial exergaming consoles, such as the Xbox system (including Xbox One and Xbox 360) and Nintendo Will (Wii Sports and Wii Fit), are available. Ogawa et al systematically reviewed 7 clinical trials (5 RCTs and 2 uncontrolled studies) and revealed that exergaming could improve cognitive functions, including executive function, process speed and reaction time, of older people. Moreover, a recent RCT revealed that, compared with the combined use of exercise (resistance, aerobic and balance training), a 12 week Kinect-based exergaming could better improve the global cognition [F(1, 44) = 5.277, p = 0.026] as measured by the Montreal Cognitive Assessment of community-frail older people. The Kinect-based group (n = 25) also demonstrated significant improvement in verbal (p < 0.05) and working (p < 0.05) memory post-intervention but the combined exercise group (n = 21) did not.

Given that sacropenia and impaired cognitive function are 2 major contributors to frailty; and exergaming and resistance training are effective treatments in improving the cognitive function and sacropenia of older people respectively, this study aims to evaluate the effects of the combined use of exergaming and resistance training in improving the frailty of nursing home residents.

ELIGIBILITY:
Inclusion Criteria:

* living in a nursing home
* fulfilled 1, 2 or 3 Fried Criteria of frailty
* score ≥7 of 10 on the Chinese version of the Abbreviated Mental Test
* able to follow the instructions of assessment and intervention

Exclusion Criteria:

* involved in any drug or other clinical trials
* having any additional medical conditions (such as epilepsy)
* unable to walk independently without the use of walking aids
* having any other conditions that will hinder the assessment and intervention (e.g.,visual/audio impairment could not be corrected by glasses/hearing aids etc).

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Muscle quantity, higher score means better muscle quantity | T1: baseline (before the study begins)
  Will be assessed using a bioelectrical impedance measurement
Change from baseline muscle quantity at 6 weeks, higher score means better muscle quantity | T2: mid-intervention (week 6)
  Will be assessed using a bioelectrical impedance measurement
Change from baseline muscle quantity at 12 weeks, higher score means better muscle quantity | T3: post-intervention (week 12)
  Will be assessed using a bioelectrical impedance measurement
Change from baseline muscle quantity at 16 weeks, higher score means better muscle quantity | T4: 1 month follow up (week 16)
  Will be assssed using a bioelectrical impedance measurement
Change from baseline muscle quantity at 24 weeks, higher score means better muscle quantity | T5: 3 months follow up (week 24)
  Will be assssed using a bioelectrical impedance measurement
Muscle strength, higher score means better muscle strength | T1: baseline (before the study begins)
  Will be assessed using a handheld dynamometer
Change from baseline muscle strength at 6 weeks, higher score means better muscle strength | T2: mid-intervention (week 6)
  Will be assessed using a handheld dynamometer
Change from baseline muscle strength at 12 weeks, higher score means better muscle strength | T3: post-intervention (week 12)
  Will be assessed using a handheld dynamometer
Change from baseline muscle strength at 16 weeks, higher score means better muscle strength | T4: 1 month follow up (week 16)
  Will be assessed using a handheld dynamometer
Change from baseline muscle strength at 24 weeks, higher score means better muscle strength | T5: 3 months follow up (week 24)
  Will be assessed using a handheld dynamometer
Lower Extremity functions, score ranged from 0-12, higher scores mean better lower extremity functions | T1: baseline (before the study begins)
  Will be assessed using the Short Physical Performance Battery
Change from baseline lower extremity functions at 6 weeks, score ranged from 0-12, higher scores mean better lower extremity functions | T2: mid-intervention (week 6)
  Will be assessed using the Short Physical Performance Battery
Change from baseline lower extremity functions at 12 weeks, score ranged from 0-12, higher scores mean better lower extremity functions | T3: post-intervention (week 12)
  Will be assessed using the Short Physical Performance Battery
Change from baseline lower extremity functions at 16 weeks, score ranged from 0-12, higher scores mean better lower extremity functions | T4: 1 month follow up (week 16)
  Will be assessed using the Short Physical Performance Battery
Change from baseline lower extremity functions at 24 weeks, score ranged from 0-12, higher scores mean better lower extremity functions | T5: 3 months follow up (week 24)
  Will be assessed using the Short Physical Performance Battery

SECONDARY OUTCOMES:
Cognitive function, higher score means better cognitive function, score ranged from 0 - 30, higher scores mean better cognition | T1: baseline (before the study begins)
  Will be assessed using the Montreal Cognitive Assessment (HK version)
Change from baseline cognitive function at 6 weeks, higher score means better cognitive function, score ranged from 0 - 30, higher scores mean better cognition | T2: mid-intervention (week 6)
  Will be assessed using the Montreal Cognitive Assessment (HK version)
Change from baseline cognitive function at 12 weeks, higher score means better cognitive function, score ranged from 0 - 30, higher scores mean better cognition | T3: post-intervention (week 12)
  Will be assessed using the Montreal Cognitive Assessment (HK version)
Change from baseline cognitive function at 16 weeks, higher score means better cognitive function, score ranged from 0 - 30, higher scores mean better cognition | T4: 1 month follow up (week 16)
  Will be assessed using the Montreal Cognitive Assessment (HK version)
Change from baseline cognitive function at 24 weeks, higher score means better cognitive function, score ranged from 0 - 30, higher scores mean better cognition | T5: 3 months follow up (week 24)
  Will be assessed using the Montreal Cognitive Assessment (HK version)
Mobility, longer time means worse functional mobility | T1: baseline (before the study begins)
  Will be assessed using the Timed Up and Go Test
Change from baseline mobility at 6 weeks, longer time means worse functional mobility | T2: mid-intervention (week 6)
  Will be assessed using the Timed Up and Go Test
Change from baseline mobility at 12 weeks, longer time means worse functional mobility | T3: post-intervention (week 12)
  Will be assessed using the Timed Up and Go Test
Change from baseline mobility at 16 weeks, longer time means worse functional mobility | T4: 1 month follow up (week 16)
  Will be assessed using the Timed Up and Go Test
Change from baseline mobility at 24 weeks, longer time means worse functional mobility | T5: 3 months follow up (week 24)
  Will be assessed using the Timed Up and Go Test
Frailty, score range 0 to 9, higher score means higher level of frailty | T1: baseline (before the study begins)
  Will be assessed using the Chinese version of Clinical Frailty Scale (CFS-C)
Change from baseline frailty at 6 weeks, score range 0 to 9, higher score means higher level of frailty | T2: mid-intervention (week 6)
  Will be assessed using the Chinese version of Clinical Frailty Scale (CFS-C)
Change from baseline frailty at 12 weeks, score range 0 to 9, higher score means higher level of frailty | T3: post-intervention (week 12)
  Will be assessed using the Chinese version of Clinical Frailty Scale (CFS-C)
Change from baseline frailty at 16 weeks, score range 0 to 9, higher score means higher level of frailty | T4: 1 month follow up (week 16)
  Will be assessed using the Chinese version of Clinical Frailty Scale (CFS-C)
Change from baseline frailty at 24 weeks, score range 0 to 9, higher score means higher level of frailty | T5: 3 months follow up (week 24)
  Will be assessed using the Chinese version of Clinical Frailty Scale (CFS-C)
Sarcopenia, score ranged from 0 to 20, lower score means lower risk | T1: baseline (before the study begins)
  Will be assessed using the Strength, Assistance with walking, Rise from a chair, Climb stairs and (Calf) Falls(SARC-Calf)
Change from baseline sarcopenia at 6 weeks, score ranged from 0 to 20, lower score means lower risk | T2: mid-intervention (week 6)
  Will be assessed using the Strength, Assistance with walking, Rise from a chair, Climb stairs and (Calf) Falls (SARC-Calf)
Change from baseline sarcopenia at 12 weeks, score ranged from 0 to 20, lower score means lower risk | T3: post-intervention (week 12)
  Will be assessed using the Strength, Assistance with walking, Rise from a chair, Climb stairs and (Calf) Falls(SARC-Calf)
Change from baseline sarcopenia at 16 weeks, score ranged from 0 to 20, lower score means lower risk | T4: 1 month follow up (week 16)
  Will be assessed using the Strength, Assistance with walking, Rise from a chair, Climb stairs and (Calf) Falls (SARC-Calf)
Change from baseline sarcopenia at 24 weeks, score ranged from 0 to 20, lower score means lower risk | T5: 3 month follow up (week 16)
  Will be assessed using the Strength, Assistance with walking, Rise from a chair, Climb stairs and (Calf) Falls (SARC-Calf)

CONTACTS AND LOCATIONS:
Locations (1):
- Jockey club Institute of Health, Ho Man Tin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The datasets of the study will only be available from the corresponding author on reasonable request after the findings being published in peer-reviewed journal.